CLINICAL TRIAL: NCT02312648
Title: Impact of an Early Mobilization Program on Functional Capacity After Coronary Artery Bypass Surgery: a Protocol of Randomized Controlled Trial.
Brief Title: Impact of Mobilization on Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luciana Chiavegato (Other)
Responsible Party: Sponsor-Investigator, Luciana Chiavegato, Professor of Master's and Doctoral Programs in Physical Therapy of Universidade Cidade de São Paulo, Universidade Cidade de Sao Paulo
Organization: Universidade Cidade de Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UNICID
Record Dates: First submitted 2014-11-08; First posted 2014-12-09 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Postoperative; Dysfunction Following Cardiac Surgery
Keywords: Functional Capacity; Physical Exertion; Patient Care; Early mobilization
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early mobilization Group (Active Comparator): Patients will perform deep breaths (3 sets of 10 repetitions), once a day, for 30 minutes until 7th postoperative day. Non invasive ventilation will be installed after orotracheal extubation for 30 to 60 minutes.Early mobilization protocol consist of upper and lower (cycle ergometer) limb exercises, chair transfer, deambulation for 10 to 20 minutes, step exercise (six times).
  Interventions: Other: Interventional Group
- Control Group - Respiratory exercise (Other): Respiratory exercises with patient sitting in bed with a high headboard 45, the same breathing exercises will be held
  Interventions: Other: Control group

INTERVENTIONS:
Other: Interventional Group — Respiratory exercises will be performed and subsequently active upper limb exercises will be conducted (flexion-extension and adduction-abduction) of large joints (shoulder, elbow and wrist) Associated with upper limb exercises, patients will undergo a series of exercises ergometer with lower limb (LL). The mobilization will be conducted on a cycle ergometer in an active, lasting 20 minutes, divided into three steps: heat 5 minutes; 10 minutes of low intensity exercise, with a speed of 30 revolutions per minute (rpm); and 5 minutes recovery. The patient remains in the supine position with the head of the bed elevated to 45 degrees, while the lower limbs will remain planned. After positioning the patient, the ergometer is adjusted.
  Arms: Early mobilization Group
Other: Control group — The patients will oriented to maintain sitting position and perform deep breaths (3 sets of 10 repetitions) in each session. They will receive the intervention once a day, for 30 minutes until 7th postoperative day. In addition, non invasive ventilation will be installed after orotracheal extubation for 30 to 60 minutes.
  Arms: Control Group - Respiratory exercise

SUMMARY:
The objective of this study is to investigate the effects of a program of early mobilization in the functional capacity in patients undergoing coronary artery bypass grafting in short and long- term.

DETAILED DESCRIPTION:
The hypotheses this study is that patients if conduct the program of early mobilization during hospitalization achieve better performance in the walk test (distance) at hospital discharge and 60 days after the surgical procedure compared to patients who only carry out the program of respiratory exercises. Intervention and control groups will receive breathing exercises up to 24 hours postoperatively, and the intervention group will also receive early mobilization exercises.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients admitted to elective and conventional coronary artery bypass, Body Mass Index (BMI) between 20 and 30 Kg/m2, mechanical ventilation time under than 24 hours, hemodynamic stability with or without use of positive inotropes, absence of arrhythmias and angina, mean arterial pressure (MAP) 60<PAM<100 mmHg, heart frequency (HR) 60<FC<100 bpm without signs of respiratory distress such as flaring nose, use of accessory muscles, thoracoabdominal asynchrony, respiratory frequency (f) ≤ 20 bpm without signs of infection were included in this study.

Exclusion Criteria:

* : presence of previous pulmonary disease, ejection fraction under 35% or longer than 54%, reoperation, intraoperative death or any contraindications to perform the proposed measurements and/or treatment.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Functional Capacity | All patients will be evaluated on preoperative period ( when they arrived in the hospital to do the surgery), hospital discharge ( about a mean of two weeks afeter surgery) and 60 postoperative days in cargiology ambulatory
  Patients will be submitted to six minute walking test

SECONDARY OUTCOMES:
Intensive Care Unit (ICU) and Hospital length of stay | All patients will be followed for the duration of hospital stay, an expected average of 30 days
  The number the days in ICU and hospital until discharge will be counted for each patient
Postoperative pulmonary complication (PPC) | All patients will be followed for the duration of hospital stay, an expected average of 30 days
  The occurrence of PPC will be monitored until the day of hospital discharge by a physician blinded to the groups: pneumonia (chest radiography with pulmonary infiltrate associated with two of the following signs: purulent expectoration, temperature above 38.3º C and a greater than 25% increase in baseline leukocyte count with hyperthermia), atelectasis (RS associated with abnormal chest acute respiratory symptoms), hypoxemia (peripheral oxygen saturation associated with respiratory symptoms below 85%).

CONTACTS AND LOCATIONS:
Overall Officials: Luciana D Chiavegato, PhD, Study Director — Universidade Cidade de São Paulo